CLINICAL TRIAL: NCT04782609
Title: A Phase 1b Dose Escalation/Dose Expansion Study of Icapamespib (PU-AD) in Patients With Recurrent Malignant Glioma
Brief Title: Study of Icapamespib (PU-AD) in Patients With Recurrent Malignant Glioma
Acronym: Glio
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Samus Therapeutics Company Closure
Sponsor: Samus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PU-AD-SD-0104
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Glioblastoma Multiforme (GBM); Grade 3 Isocitrate Dehydrogenase (IDH) Wildtype Astrocytoma; Grade 3 or 4 Astrocytoma; Glioblastoma Surgery
MeSH Terms: conditions — Glioblastoma; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Part 1 of the trial will be a standard 3 by 3 dose escalation design where different doses are examined. Part 2 will be a dose expansion cohort to further evaluate the recommended Phase 2 dose (RP2D). The RP2D is defined as the dose level recommended for further clinical study, or the highest dose tested. The RP2D may be the same as the MTD or modified from the MTD based on assessment of overall exposure, safety experience in Cycle 2 and beyond, and clinical benefit data in the study. The RP2D will be determined in the dose expansion phase of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20 mg Icapamespib cohort (Experimental): Icapamespib will be administered orally once daily for each 28-day cycle. The initial dose in this trial will be 20 mg
  Interventions: Drug: Icapamespib
- dose expansion cohort (Experimental): dose expansion cohort to further evaluate the recommended Phase 2 dose (RP2D)
  Interventions: Drug: Icapamespib

INTERVENTIONS:
Drug: Icapamespib — to test the safety, tolerability and pharmacokinetics of single agent oral icapamespib in patients with recurrent brain lesions.
  Other Names: Malignant Glioma

SUMMARY:
This is a 2-part multicenter Phase 1b study designed to test icapamespib in patients with recurrent brain lesions.

Part 1 of the trial will be a standard 3 by 3 dose escalation design where different doses are examined. Part 2 will be a dose expansion cohort to further evaluate the recommended Phase 2 dose (RP2D). The RP2D is defined as the dose level recommended for further clinical study, or the highest dose tested.

DETAILED DESCRIPTION:
This is a 2-part multicenter Phase 1b study designed to test the safety, tolerability and pharmacokinetics of single agent oral icapamespib in patients with recurrent brain lesions.

Part 1 of the trial will be a standard 3 by 3 dose escalation design where different doses are examined. Part 2 will be a dose expansion cohort to further evaluate the recommended Phase 2 dose (RP2D). The RP2D is defined as the dose level recommended for further clinical study, or the highest dose tested. The RP2D may be the same as the maximum tolerated dose (MTD) or modified from the MTD based on assessment of overall exposure, safety experience in Cycle 2 and beyond, and clinical benefit data in the study. The RP2D will be determined in the dose expansion phase of the study.

Part 1: Up to 30 patients with 1st, 2nd or 3rd recurrence of IDH wild type glioblastoma multiforme (GBM) or grade 3 or 4, Isocitrate dehydrogenase (IDH) mutant astrocytoma will be enrolled to evaluate the safety, pharmacokinetics (PK), pharmacodynamics, and MTD of single agent oral icapamespib administered daily.

Icapamespib will be administered orally once daily for each 28-day cycle. The initial dose in this trial will be 20 mg in Cohort 1. Dose escalation will proceed as follows:

* 100% increment until the first drug-related Grade 2 adverse event (AE) occurs, then
* 50% increment until the first drug-related Grade 3 event occurs, then
* 33% increment until the first Dose Limiting Toxicities (DLT) occurs, then
* 20% increment until RP2D is declared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects having histologically confirmed IDH wildtype glioblastoma (Parts 1 and 2), or grade 3 or 4 IDH mutant astrocytoma (Part 1 only) per WHO criteria
* Subjects must be at 1st, 2nd, or 3rd recurrence (Part 1) or 1st or 2nd recurrence (Part 2) and with at least 5 subjects clinically requiring reoperation for tumor progression (Part 2). ; Note: recurrence is defined as progression following initial therapy (i.e., radiation, chemotherapy, or radiation + chemotherapy); if the participant had a surgical resection for relapsed disease and no anti-tumor therapy instituted for up to 12 weeks, this is considered one recurrence.
* Measurable disease as defined by modified RANO (1 cm × 1 cm minimum dimensions, at least 12 weeks after final radiotherapy dose; if new disease is outside radiotherapy field, <4 weeks is acceptable).
* Cranial MRI performed within 14 days prior to study entry.
* Age equal to or greater than 18 years
* Karnofsky performance status of >60 at screening
* Adequate bone marrow, liver and renal functions (tests must be performed within 14 days prior to enrollment).The following laboratory values must be documented within 3 days prior to the first dose of study drug Absolute neutrophil count (ANC) ≥1.5 × 109/L Platelet count ≥100 × 109/L Estimated creatinine clearance (CrCl) >60 mL/min by Cockcroft-Gault formulation Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 × the upper limit of normal (ULN) Total bilirubin ≤1.5 × ULN (unless due to Gilbert's syndrome) Serum albumin ≥2.8 g/dL International normalized ratio (INR) <1.5 (except subjects maintained on anticoagulant medications)
* Negative serum or urine pregnancy test (females of childbearing potential only).
* Willingness to follow highly effective means of contraception
* Able and willing to give informed consent

Exclusion Criteria:

* Currently receiving any concomitant anti-cancer medication
* Prior treatment with Gliadel wafers.
* No radiation within 4 weeks of starting treatment.
* Has tumor localized primarily to the brainstem or spinal cord.
* A history of any other primary malignancy that has not been treated with curative intent and that has not been in complete remission for at least 2 years (exempt from the two year limit are non-melanoma skin cancer and cervical carcinoma in-situ on biopsy or a squamous intraepithelial lesion on PAP smear).
* Active infection requiring systemic treatment.
* Any significant medical illnesses or toxicities that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy. Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism, e.g. congestive heart failure, moderate to severe liver and renal disease, other cancers.
* History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class III or IV) or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to Screening
* QT interval corrected with the Fridericia formula (QTcF) on average of triplicate ECG readings (taken approximately 5 minutes apart) at Screening Visit ECG or Baseline Visit ECGs >450 msec for males or >470 msec for females (except when QT prolongation is associated with right or left bundle branch block, in which case enrollment is allowed).
* Has active ocular condition unrelated to primary intracranial pathology, that in the opinion of the investigator, may alter visual acuity during the course of the study.
* The need for concomitant use of long-acting gastric pH elevating agents (proton pump inhibitors or H2-receptor antagonists) at study entry and during the study (note: gastric locally-acting antacids may be allowed if administered >2 hours before or after dosing).
* The need for concomitant use of any drugs that are sensitive substrates of CYP 450 isozymes with narrow therapeutic index for at least 7 days prior to administration of the first dose of IMP and throughout the study.
* The need for concomitant use of any drugs that are strong inhibitors or inducers of cytochrome (CYP) 450 isozymes at least 7 days prior to administration of the first dose of IMP and throughout the study.
* Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug, whichever is longer, prior to first dose of IMP in this study; or is currently participating in another clinical study.
* Has taken corticosteroids at greater than dexamethasone 4 mg daily or equivalent daily, participants taking <4 mg daily are eligible if the dose has been stable for ≥ 1 week before the first dose of study drug.
* Other unspecified reasons that, in the opinion of the investigator or Samus and/or its delegated medical monitor, place the subject at risk or make the subject unsuitable for the study or unable or unwilling to comply with the requirements of the study
* History or presence of conditions, which in the judgment of the investigator, are known to interfere with the absorption distribution, metabolism or excretion of drugs, such as prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy)
* Prior exposure to icapamespib or other Hsp90 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5
Maximum Tolerated Dose (MTD)/Coverage with evidence development (CED)/recommended phase 2 dose (RP2D) (Part 1 Only | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  Assessed by the occurrences of DLTs in doses of single agent icapamespib. The MTD will be defined as the dose that does not exceed an acceptable threshold of toxicity which is set at 33%. Scientific Review Committee (SRC) may elect to set the dose lower than MTD or in the absence of establishing MTD as the Recommended Phase 2 dose (RP2D).
Icapamespib Plasma Concentration at Time of Surgery | 7-14 days post surgery
  Tissue samples collected at surgery after icapamespib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD, Study Director — Samus Therapeutics
Locations (5):
- United States (5):
  - University of California, Las Angeles Medical Center, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No